CLINICAL TRIAL: NCT02688010
Title: Effect of Reduced Noise Levels and Cycled Light on Visual and Neural Development in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CHFudanU_NNICU7
Record Dates: First submitted 2016-01-30; First posted 2016-02-23 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Preterm Infants
Keywords: noise; sound; cycled light; preterm infants; neonatal care; growth; visual development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No specific noise reduction strategies to restrict noise exposure less than 45 dB combined with either continuous bright light or continuous near darkness or unstructured combination of the two during the hospitalization.
- Noise reduction and cycled light (Experimental): Reduced noise exposure (sound levels <45 dB) and cycled light (approximately 12 hours of light on and 12 hours of light off).
  Interventions: Behavioral: Noise reduction and cycled light

INTERVENTIONS:
Behavioral: Noise reduction and cycled light — Reduced noise exposure (sound levels <45 dB) and cycled light (approximately 12 hours of light on and 12 hours of light off).
  Arms: Noise reduction and cycled light

SUMMARY:
Noise is a hazard for newborn. In 1997, the American Academy of Pediatrics determined that safe sound levels in the neonatal intensive care unit (NICU) should not exceed 45 dB which has been rarely achieved. High intensities of noise have several negative effects on preterm newborns. Also, they are exposed to either continuous bright light continuous near darkness or unstructured combination of the two during their hospitalizations. The investigators primary objective is to determine the impact of reduced noise levels and cycled light on growth parameters and visual development in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* <37 gestational weeks preterm infants and >1250g birth weight

Exclusion Criteria:

* Major congenital anomaly and infection prior to enrolment
* Infants with surgical issues

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Flash visual evoked potentials (FVEP) at 4 weeks of age | at 4 weeks of age
  FVEP is recorded from each eye individually after they fall asleep. Three silver-sliver chloride electrodes are placed according to 10-20 International system with active electrode at Oz (1-2 cm above inion), reference electrode at Fz and ground electrode at Cz. Scalp-electrode impedance is usually below 5kΩ but always below 10kΩ. Flash stimulus (2 Hz.) is given by light emitting diode goggles simulator at a distance of 2 cm to one eye at a time. 100 responses are averaged for each eye automatically in the Nicolet Viking Quest visual electrophysiological device at 1s total sweep time. Band pass filters are set at 0.1-75 Hz. The reproducibility of the responses is ensured by repeating the test two or more times. Responses with excessive artifacts are automatically rejected. The parameters of P1, N1, P2, N2, P3, and N3 of the FVEP are stored and subsequently assessed by ophthalmologist blinded to the infant's clinical course.
Bayley Scales of Infant Development, Second Edition (BSID-III) at 18 months of age | at 18 months of age
  Neurodevelopment outcome is measured with the Bayley Scales of Infant Development, Second Edition (BSID-III) at corrected gestational age of 18 month, assessed by the physician from department of child health care who was blinded with respect to the subjects. Mental and motor scores were calculated by the BSID-III Mental Developmental Index (MDI) and Psychomotor Developmental Index (PDI). The subject's neurodevelopmental outcome was classified as delayed if either score was less than 70.

SECONDARY OUTCOMES:
Time to establish full enteral feeding | birth till discharge from hospital (up to 3 months)
  up to 3 months
Weight at discharge | birth till discharge from hospital (up to 3 months)
  up to 3 months
Head circumferences at discharge | up to 3 months
Incidence of nosocomial infection | up to 3 months
Incidence of retinopathy of prematurity | up to 3 months
Incidence of intraventricular hemorrhage | 1 month
Incidence of bronchopulmonary dysplasia | at corrected gestational age of 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Dr., Study Chair — Key Laboratory of Neonatal Diseases, Ministry of Health
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Noise: a hazard for the fetus and newborn. American Academy of Pediatrics. Committee on Environmental Health. Pediatrics. 1997 Oct;100(4):724-7. No abstract available. PMID 9836852
- [Result] Lasky RE, Williams AL. Noise and light exposures for extremely low birth weight newborns during their stay in the neonatal intensive care unit. Pediatrics. 2009 Feb;123(2):540-6. doi: 10.1542/peds.2007-3418. PMID 19171620
- [Result] Laudert S, Liu WF, Blackington S, Perkins B, Martin S, Macmillan-York E, Graven S, Handyside J; NIC/Q 2005 Physical Environment Exploratory Group. Implementing potentially better practices to support the neurodevelopment of infants in the NICU. J Perinatol. 2007 Dec;27 Suppl 2:S75-93. doi: 10.1038/sj.jp.7211843. PMID 18034183
- [Result] Morag I, Ohlsson A. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2013 Aug 3;(8):CD006982. doi: 10.1002/14651858.CD006982.pub3. PMID 23913547
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174